CLINICAL TRIAL: NCT00144144
Title: A Randomized, Controlled Study on Calcium Channel Blocker Versus Angiotensin II Antagonists in the Hypertensive Patients With Type 2 Diabetes Mellitus Under the Inadequately Controlled Blood Pressure With Angiotension II Antagonists
Brief Title: A Study on Ca Blocker Versus AII Antagonists in Hypertension With Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Advanced-J (Other)
Collaborators: Japan Heart Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADVANCED-J01; UMIN-C000000017
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2006-07-14 (Estimated); Status verified 2006-07

CONDITIONS: Hypertension; Diabetes Mellitus, Type 2
Keywords: Hypertension; Diabetes Mellitus, Type 2; Calcium Channel Blocker; Angiotensin II type 1 Receptor Blocker
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — Angiotensin Receptor Antagonists; Calcium Channel Blockers

INTERVENTIONS:
Drug: Angiotensin II receptor antagonists, Calcium channel blocker

SUMMARY:
The antihypertensive effect of the increased dose of angiotensin II receptor blocker (AII antagonist) is compared with that of the additional combined use of amlodipine in hypertensive patients with Type 2 diabetes mellitus, who have been treated with AII antagonist, the antihypertensive effect of which has been inadequate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus.
* Patients who have been treated by the single use of AII antagonist at usual for at least 8 weeks or patients who have been treated by the combined use of AII antagonist at usual doses and calcium channel blocker or a antihypertensive drug other than ACE inhibitors for at least 8 weeks.
* Patients who show a systolic blood pressure (blood pressure) > 135 mm Hg or a diastolic blood pressure > 85 mm Hg, which is measured (in a sitting position) on an outpatient basis at the time of start of the observation period, and show the mean (blood pressure level measured at home after getting up before the start of study) of systolic blood pressure > 130 mm Hg or diastolic blood pressure > 80 mm Hg measured at home after getting up for last 5 days during the last 2-week observation period.
* Patients whose consent is obtained at age 20 years or over.
* Patients whose consent is obtained from themselves in written form. With regard to 2) and 3), however, the case, in which the mean of the systolic blood pressure levels measured at home after getting up for last 5 days during the first 1-week observation period is > 180 mm Hg or the mean diastolic blood pressure level is > 110 mm Hg, is included in the present study.

Exclusion Criteria:

* Patients with secondary hypertension.
* Patients who show a systolic blood pressure > 180 mm Hg or diastolic blood pressure > 110 mm Hg on the measurement (in a sitting position) on an outpatient basis at the time of start of the observation period.
* Patients with severe hepatic dysfunction.
* Patients with severe renal dysfunction.
* Patients with a past history of hypersensitiveness to study drugs.
* Pregnant, lactating, and probably pregnant patients, and patients who want to become pregnant during the study period.
* Patients who have participated in the trial within 3 months before the start of the observation period or who attend the trial simultaneously with the present study.
* Other patients judged as being inappropriate for the subjects of the study by investigators.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-09; Study Completion 2008-09

PRIMARY OUTCOMES:
Changes in blood pressure level at home after getting up.
The rate of the blood pressure levels at home after getting up, which effected the target levels (systolic blood pressure < 125 mm Hg, diastolic blood pressure < 80 mm Hg).
Adverse events, adverse drug reactions
Clinical laboratory data

SECONDARY OUTCOMES:
Changes in blood pressure levels measured on an outpatient basis.
The rate of the blood pressure levels measured on an outpatient basis, which effected the standard levels (systolic blood pressure level <130 mm Hg, diastolic blood pressure level < 80 mm Hg).
Changes in blood pressure levels measured at home before going to bed· Changes in IMT of the cervical artery
Changes in PWV· Changes in echocardiographic findings
Changes in urinary albumin level
Changes in BNP· Changes in hs-CRP· Medical cost-effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Ryuzo Kawamori, M.D., Principal Investigator — Juntendo University School of Medicine, Dept. of Endocrinology and Metabolism
Locations (1):
- Dept. of Clinical Immunology, Clinical Bioinformatics Research Unit, Graduate School of Medicine, the University of Tokyo, Hongo, Bunkyo-ku, Tokyo, Japan